CLINICAL TRIAL: NCT03994835
Title: 2000 HIV Human Functional Genomics Partnership Program
Acronym: 2000HIV
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: ViiV Healthcare (Industry); Elisabeth-TweeSteden Ziekenhuis (Other); Erasmus Medical Center (Other); Onze Lieve Vrouwe Gasthuis (Other)
Responsible Party: Sponsor
Other Study IDs: NL.68056.091.18
Record Dates: First submitted 2019-05-22; First posted 2019-06-21 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: HIV Infections
Keywords: HIV; Non-alcoholic fatty liver disease; Cardiovascular disease; Omics data; Inflammation
MeSH Terms: conditions — HIV Infections; Non-alcoholic Fatty Liver Disease; Cardiovascular Diseases; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood for DNA isolation (no sequencing, only SNP array) Stool for microbiome analysis Saliva for microbiome analysis Plasma and serum for metabolomics Urine for creatinine analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background Chronic HIV infection leads to a dysregulated immune system, even when full viral suppression is achieved. HIV causes persistent immune activation, relating to an array of common non-AIDS-related diseases such as cardiovascular disease (CVD) and non-alcoholic fatty liver disease (NAFLD). On the other hand, accelerated ageing of the immune system hinders effective immunity against infectious diseases and cancer. Likewise, this derailed inflammatory balance creates a niche for persistent viral replication and reservoir, and prevents cure or functional cure. Mechanisms behind this phenomenon are poorly understood. Inclusion of a larger cohort of HIV-infected patients allows for a more precise assessment of the factors underlying the immune dysregulation.

Primary Objectives

* Identify a set of candidate biomarkers that correlate with particular non-AIDS-related comorbidities
* Unravel biological processes associated with extreme HIV clinical phenotypes.
* Find therapeutic targets to identify novel assets or for repurposing of clinical phase assets from other disease areas for HIV.

Secondary Objectives

* Evaluate potential relationship of host/immune profiles on efficacy, safety, and tolerability of standard care regimens.
* Evaluate the contribution of age, sex, and genetics in host-immune profiles that are:

  * distinct to HIV infection relative to controls in other cohorts;
  * associated with non-AIDS-related comorbidities in HIV infection relative to non-HIV chronic disease.

Study design 2000 HIV patients will be included in the cohort. The investigators estimate a 2-year inclusion and 2-year follow-up period and will strive for the inclusion of several clinical phenotypes and classical risk group patients. Patients will be recruited from four Dutch HIV treatment centers.

At inclusion

1. Collection of metadata using questionnaires and patient medical records
2. Asses co-pathology (CVD and NAFLD)
3. Blood will be drawn for genetic, epigenetic, proteomic, metabolomic, microbiome, immunological, and virological analyses

After 2 years follow-up

1. Collection of metadata using questionnaires and patient medical records
2. Asses co-pathology (CVD and NAFLD)
3. Blood samples will be collected for biomarker and infection/inflammation parameter analysis

DETAILED DESCRIPTION:
Study population A cohort with a total of 2000 HIV patients will be built, consisting of a discovery cohort (n=1200) and confirmation cohort (n=800). The investigators estimate a 2-year inclusion and 2-year follow-up period and will strive for the inclusion of several clinical phenotypes such as long-term non-progressors (~2-3%), immunologic non-responders (~3%), and rapid progressors (~4-5%) and classical risk group patients such as men who have sex with men (MSM), females, and subjects from Sub-Sahara Africa. Patients will be recruited from the following Dutch HIV Treatment Centers: Radboudumc (Nijmegen), Erasmus MC (Rotterdam), OLVG (Amsterdam), Elisabeth Twee-Steden Ziekenhuis (Tilburg).

A sample size calculation cannot be provided due to the variable frequencies of the various traits in genome-microbiome interaction, and their effect on cytokine production. Because of the explorative nature of this study, the size calculation will be variable depending on the type of polymorphism analyzed. The frequencies of the various microorganism classes in the colonizing microbiome is not known in our study population, and therefore power calculations are impossible to be performed.

Earlier studies in the Human Functional Genomics Project have assessed microbiome traits in 250-500 individuals. An earlier HFGP study included a uniform cohort of 200 HIV-infected individuals (all MSM). The present study will also include HIV-infected patients with a more extreme phenotype, females and subjects originating from Sub-Sahara Africa. Because of this, the investigators decided to increase the number of individuals tested to 2000, consisting of a discovery cohort of 1200 subjects, and a confirmation cohort of 800 participants.

Study visits and procedures At inclusion

1. The investigators will collect metadata using questionnaires on lifestyle, health and clinical symptoms, including neuropsychiatric symptoms. Relevant data will also be collected from the patients records in the medical centers and the HIV Monitoring Foundation.
2. Co-pathology will be assesed:

   * Cardiovascular risk scores (D:A:D risk score and Framingham CVD score) will be collected as well as ECG and intima-media thickness (IMT) measurements.
   * Non-Alcoholic Fatty Liver Disease (NAFLD) assessment through liver ultrasound and FibroScan.
3. Blood will be drawn (90 ml):

   * DNA will be isolated for genetic and epigenetic analysis.
   * The function of the immune system will be analyzed at several levels using circulating white blood cells from venous blood.
   * Metabolism and proteomics will be analyzed
   * Virological analysis, characterizing the HIV reservoir, HIV resistance and viral sequences in circulating DNA and RNA.
4. Microbiome analysis will be performed on stool and saliva samples.
5. Urine sample will be collected for creatinine measurements and microbiome.

After 2 years follow-up

1. The investigators will collect metadata using questionnaires on lifestyle, health and clinical symptoms, including neuropsychiatric symptoms. Relevant data will also be collected from the patients records in the medical centers and the HIV Monitoring Foundation.
2. Co-pathology will be assesed:

   * Cardiovascular risk scores (D:A:D risk score and Framingham CVD score) will be collected as well as ECG.
   * Non-Alcoholic Fatty Liver Disease (NAFLD) assessment through liver ultrasound and FibroScan.
3. Blood samples (10ml) will be collected for biomarker and infection/inflammation parameter analysis.

Patient informed consent procedure Patients will always be approached first by a treating physician or specialized nurse. They will be provided with information and will be asked if a physician-researcher may contact the patient. If there is oral consent for this, the researcher contacts the patient in one week to ask if they are interested in participating in the study. the physician-researcher will answer any questions the patient may have and plan the first visit. The informed consent procedure will be conducted during the patient's first visit.

Patient registry procedures All patient data will be recorded only in coded form in a secure database with audit and edit trail (CASTOR EDC). During the informed consent procedure, the patient is given a study code. The identifying patient data and study code is kept in a password-protected key file, only accessible to the local research team. No patient-identifying data will leave the local medical center.

In the questionnaires and eCRFs in CASTOR, the investigators will enter as many data checks as possible

Biomaterials All biomaterial (blood, stool, urine, saliva) will be transported to and processed in the laboratory of Experimental Internal Medicine of the Radboudumc in Nijmegen. Here, all the biomaterial will also be stored collectively. All materials will be handled and stored only under the patient's study code.

Monitoring Monitoring will be performed by an independent monitor according to the latest guidelines of the The Netherlands Federation of University Medical Centers. An initiation and close-out visit will be planned in plenary form with all the centers in Radboudumc. There will be one extra visit per center. During these visits informed consents will be checked, as well as inclusion and exclusion criteria and source data verification in a small subset of total participants.

Data collection for patient registry

Baseline data collected from electronic patient files or the HIV Monitoring Foundation during inclusion visit:

Medical history:

1. Inclusion date
2. Length and weight
3. Last known blood pressure (and date measured)
4. Seroconversion date (if known)
5. Date first HIV-positive test
6. Date start cART
7. HIV transmission risk behavior:

   * MSM
   * Heterosexual
   * Injecting drug use
   * Contaminated blood products
   * Unknown
8. First CD4 count
9. CD4 nadir
10. CD4/CD8 ratio pre-cART
11. HIV stadium at start cART according to CDC criteria
12. Pre-cART HIV RNA zenith
13. Opportunistic conditions before start cART

    * None
    * MTB
    * Fungal infections
    * Parasitic infections,
    * Bacterial infections
14. Malignancies before start cART

    * None
    * If yes, specify what kind, when and treatment
15. Other known medical problems before start cART, which require long-term treatment

    * None
    * If yes, specify what kind, when and treatment
16. Response cART:

    * Period between start cART and viral load < 500 (months)
    * Viral loads:

      * Undetectable after 24 weeks: yes/no
      * Number/frequency of residual viremia (positive test with signal <50 copies): last year and last 5 years
      * Number of viral blips (50-200): last year and last 5 years
      * Number of viremia: 200-1000: last year and last 5 years
      * Number of failing cART (>1000): last year and last 5 years
      * Resistance associated mutations pre-cART and following failure
      * CD4 reconstitution
      * CD4/CD8 ratio and normalization >1 yes/no after cART initiation
17. IRIS, yes/no
18. Opportunistic conditions after start cART (if known)

    * None
    * MTB
    * Fungal infections
    * Parasitic infections,
    * Bacterial infections
19. Malignancies after start cART (if known)

    * None
    * If yes, specify what kind, when and treatment
20. Vascular diseases after start cART:

    * None
    * Stroke/ TIA
    * Angina pectoris
    * Myocardial infarction
    * Claudicatio intermittens
    * Venous thrombo-embolism
    * Other …
21. SOAs

    * None
    * HAV: yes/no, if yes: treatment and how often
    * HBV:

      * Infected: active infection (PCR+) or non-active infection
      * Vaccination: No/Yes

        * Once with anti-HBs> 100
        * Two times vaccination leading to
    * anti-HBs> 100
    * anti-HBs< 100

      * No infection
    * HCV: yes/no, if yes: treatment and how often
    * Lues: yes/ no: if yes: treatment and how often
    * Chlamydia/Go: yes/ no: if yes: treatment and how often
    * HPV
22. COVID-19 infection before or after start cART:

    * Was a COVID-19 test done and if so type of test if known (PCR or antigen test), date of test and result of laboratory test for COVID-19 (positive or negative)
    * COVID-19 Serology results
    * Register COVID-19-related hospital admissions
    * COVID-19 vaccination: type and date(s)
    * Side effects of COVID-19 vaccination:

      * Mild: overall malaise, fatigue, muscle ache, pain at injection site, shivers, headache.
      * Moderate: mild symptoms to the extend (self)medication/pain relief is required.
      * Severe: fever >38.5 degrees Celsius and/or one or more days bedridden
23. cART regimes

    * Reasons for switching
24. Prescribed co-medication
25. Full current medication list

Physical examination

* Signs of Kaposi sarcoma
* Lymphadenopathy
* For determination of medication levels: when was the last date and time HIV-medication was taken?
* Other abnormalities: …

Cardiovascular risk profile:

* D:A:D (R) and Framingham scores
* ECG

Laboratory results of date closest to inclusion date (standard care at least once a year according to Dutch guidelines):

* Full blood count
* Liver enzymes (ALAT, AF, bilirubin)
* Creatinine
* HIV-RNA
* CD4 and CD8 counts
* Glucose
* Lipid profile
* TPHA/VDRL
* HCV serology (for all at risk, such as MSM and i.v. drug users)

  * If positive, HCV PCR
* HPV diagnostics in females (PAP, PCR)
* Urine diagnostics (if available): α1-microglobulin, protein, albumin, phosphate, creatinin

Baseline data collected from electronic patient files or the HIV Monitoring Foundation during 2-year follow-up visit:

Medical history last 2 years:

1. Date of 2 year follow-up visit
2. Weight
3. Last known blood pressure (and date measured)
4. Response cART last 2 years

   * Number of residual viremia: last 2 years
   * Number of viral blips (20-200): last 2 years
   * Number of viremia (200-1000): last 2 years
   * Number of failing cART (>1000): last 2 years
   * CD4 count
   * CD4/CD8 ratio (if known)
5. Opportunistic conditions last 2 years

   * None
   * MTB
   * Fungal infections
   * Parasitic infections,
   * Bacterial infections
6. Malignancies in the last 2 years

   * None
   * If yes, specify what kind, when and treatment
7. Signs/symptoms of cardiovascular diseases in the last 2 years:

   * None
   * Stroke/ TIA
   * Angina pectoris
   * Myocardial infarction
   * Claudicatio intermittens
   * Venous thrombo-embolism
   * Other …
8. New SOAs in the last 2 years

   * HAV: yes/no, if yes: treatment and how often
   * HBV:

     * Infected: active infection (PCR+), non-active infection,
     * Vaccination: No/Yes

       * Once with anti-HBs> 100
       * Two times vaccination leading to
   * anti-HBs> 100
   * anti-HBs< 100

     * No infection
   * HCV: yes/no, if yes: treatment and how often
   * Lues: yes/ no: if yes: treatment and how often
   * Chlamydia/Go: yes/ no: if yes: treatment and how often
9. COVID-19 infection before or after start cART:

   * Was a COVID-19 test done and if so type of test if known (PCR or antigen test), date of test and result of laboratory test for COVID-19 (positive or negative)
   * COVID-19 Serology results
   * Register COVID-19-related hospital admissions
   * COVID-19 vaccination: type and date(s)
   * Side effects of COVID-19 vaccination:

     * Mild: overall malaise, fatigue, muscle ache, pain at injection site, shivers, headache.
     * Moderate: mild symptoms to the extend (self)medication/pain relief is required.
     * Severe: fever >38.5 degrees Celsius and/or one or more days bedridden
10. cART regimes in the last 2 years

    * Reasons for switching available from 'Stichting HIV Monitoring'
11. Prescribed co-medication
12. Full current medication list

Physical examination

* Signs of Kaposi sarcoma
* Lymphadenopathy
* For determination of medication levels: when was the last date and time HIV-medication was taken?
* Other abnormalities: …

Cardiovascular risk profile:

* D:A:D (R) and Framingham scores
* ECG

Laboratory results of date closest to follow-up visit date:

* Full blood count
* Liver enzymes (ALAT, AF, bilirubin)
* Creatinine
* HIV-RNA
* CD4 and CD8 counts
* Glucose
* Lipid profile
* TPHA/VDRL
* HCV serology

  o If positive, HCV PCR
* HPV diagnostics in females (PAP, PCR)
* Urine diagnostics

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected,
* aged ≥18 years,
* on cART ≥6 months with an HIV-RNA load <200 copies/mL, *Apart from the above-mentioned subjects, elite controllers that are not on cART, are also eligible.

Exclusion Criteria:

* No informed consent
* Insufficient communication because of language or other problems
* Active hepatitis B/C or signs of acute infections
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients (n=2000) will be recruited from the following Dutch HIV Treatment Centres: Radboudumc (Nijmegen), ErasmusMC (Rotterdam), Onze Lieve Vrouwe Gasthuis (Amsterdam), Elisabeth-TweeSteden Ziekenhuis (Tilburg). Our aim is to include approximately 20% females, 20% of Sub-Sahara African origin, elite controllers (~2-3%), immunologic non-responders (~3%), and rapid progressors (~4-5%) The total number of adult HIV patients under care in these treatment centers is 7000, of which 80% is male and 70% is of Caucasian origin. There is wide age distribution among the adult HIV population.
Sampling Method: Non-Probability Sample
Enrollment: 1910 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Change in liver fibrosis | Change: 2-year value - baseline value
  Change in liver fibrosis measurement by FibroScan (method by Echosens)
Change in liver steatosis | Change: 2-year value - baseline value
  Change in liver steatosis measurement by FibroScan (method by Echosens) and liver ultrasound (method developed by Radboudumc)
Change in cardiovascular risk score (Framingham score) | Change: 2-year value - baseline value
  Framingham score
Change in cardiovascular risk score (D:A:D score) | Change: 2-year value - baseline value
  D:A:D score
Number and type of cardiovascular events | Number of events over 2 years between baseline and 2-year time point
  Recoring of cadiovascular diseases from patient file:
  * Stroke/ TIA
  * Angina pectoris
  * Myocardial infarction
  * Claudicatio intermittens
  * Venous thrombo-embolism
  * Other …
Genetic data | At baseline only
  Genome-wide genotype data including >8 million SNPs per individual
Colonizing microbiome profile | At baseline only
  Colonizing microbiome profile will be generated from stool and saliva samples
Transcriptomics | At baseline only
  RNA-sequencing will be performed in PBMCs
Quantification of a wide range of metabolites | At baseline only
  Metabolomics analysis by multiplex immunoassays will be performed in plasma or serum
Cytokine production of PBMCs in ex vivo stimulation experiments | At baseline only
  Ex vivo cytokine responses of isolated PBMCs to a range of stimuli (TLR ligands, killed pathogens and viral antigen stimuli)
Immune phenotyping | At baseline only
  Extensive phenotyping of circulating immune cells by flow cytometry analysis
Change in ECG | ECG paramater changes between baseline and 2-year time visit
  Standardized signs of myocardial infarction with MEANS ECG software, as extensively described elsewehere. In addition, we will look at the full list of ECG output measurements as described elsewhere*: in brief, MEANS reliably provides output on interpretation of the ECG rhythm and morphology. The morphological interpretation consists of separate analyses of the P wave, QRS complex, and ST-T segment. Reference: Van den Berg ME, Rijnbeek PR, Niemeijer MN, et al. Normal values of corrected heart-rate variability in 10-second electrocardiograms for all ages. Front Physiol. 2018;9:424
Intima-media thickness | At baseline only
  Ultrasound measurement of intima-media thickness in the carotid artery as a measure for atherosclerosis and cardiovasculr disease risk.

CONTACTS AND LOCATIONS:
Overall Officials: Quirijn de Mast, Dr., Principal Investigator — Radboud University Medical Center; Annelies Verbon, Prof., Principal Investigator — Erasmus Medical Center; Willem Blok, Dr., Principal Investigator — Onze Lieve Vrouwe Gasthuis; Marvin Berrevoets, Drs., Principal Investigator — Elisabeth Twee-Steden ziekenhuis
Locations (4):
- Netherlands (4):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Radboudumc, Nijmegen
  - Erasmus MC, Rotterdam
  - Elisabeth Twee-Steden ziekenhuis, Tilburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Blaauw MJT, Navas A, Vasquez VR, Vadaq N, Berrevoets MAH, Otten T, Vos WAJW, van Eekeren LE, Groenendijk AL, Weijers G, Lutgens E, Koenen HJPM, de Jonge MI, Netea MG, Rutten JHW, van der Ven AJAM, Riksen NP. Functional and transcriptional senescence profiles of CD8+ T cells associate with the presence of carotid plaques in people living with HIV. J Infect Dis. 2026 Jan 7:jiag018. doi: 10.1093/infdis/jiag018. Online ahead of print. PMID 41498526
- [Derived] Blaauw MJT, Berrevoets MAH, Vos WAJW, Groenendijk AL, van Eekeren LE, Vadaq N, Weijers G, van der Ven AJAM, Rutten JHW, Riksen NP. Traditional Cardiovascular Risk Factors Are Stronger Related to Carotid Intima-Media Thickness Than to Presence of Carotid Plaques in People Living With HIV. J Am Heart Assoc. 2023 Oct 17;12(20):e030606. doi: 10.1161/JAHA.123.030606. Epub 2023 Oct 7. PMID 37804189
- [Derived] Vadaq N, Zhang Y, Vos WA, Groenendijk AL, Blaauw MJ, van Eekeren LE, Jacobs-Cleophas M, van de Wijer L, Dos Santos JC, Gasem MH, Joosten LA, Netea MG, de Mast Q, Fu J, van der Ven AJ, Matzaraki V. High-throughput proteomic analysis reveals systemic dysregulation in virally suppressed people living with HIV. JCI Insight. 2023 Jun 8;8(11):e166166. doi: 10.1172/jci.insight.166166. PMID 37079385